CLINICAL TRIAL: NCT04393038
Title: A Phase 2/3, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy and the Safety of ABX464 in Treating Inflammation and Preventing COVID-19 Associated Acute Respiratory Failure in Patients Aged ≥ 65 and Patients Aged ≥18 With at Least One Additional Risk Factor Who Are Infected With SARS-CoV-2.
Brief Title: ABX464 in Treating Inflammation and Preventing Acute Respiratory Failure in Patients With COVID-19
Acronym: Mir-Age
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interim analysis concludes that the study is futile
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABX464-401
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
Keywords: COVID-19; ABX464
MeSH Terms: conditions — COVID-19 | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Phase 2/3, randomized, double blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded treatment bottles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABX464 (Experimental): ABX464 - Capsules + Standard of Care (SOC)
  Interventions: Drug: ABX464
- Placebo (Placebo Comparator): Placebo - Capsules + Standard of Care (SOC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX464 — ABX464 50mg QD for 28 days + Standard of Care
  Arms: ABX464
Drug: Placebo — Placebo 50mg QD for 28 days + Standard of Care
  Arms: Placebo

SUMMARY:
A phase 2/3, randomized, double blind, placebo-controlled study to evaluate the efficacy and the safety of ABX464 in treating inflammation and preventing acute respiratory failure in patients aged ≥65 and patients aged ≥18 with at least one additional risk factor who are infected with SARS-CoV-2 (the MiR-AGE study).

DETAILED DESCRIPTION:
This phase 2/3 study will evaluate the efficacy and safety of ABX464 50mg QD (oral capsule), on treating inflammation and preventing acute respiratory failure in patients infected with SARS-CoV-2.

Eligible patients will be randomized according to a 2:1 ratio into 2 treatment cohorts as follows:

* Standard of Care + Placebo cohort: 344 patients
* Standard of Care + ABX464 50mg QD: 690 patients

Study design:

The study will consist of 2 periods:

* Treatment phase: randomized patients will be treated for 28 days
* Safety follow-up phase of 14 days after which the End of Study visit (EOS) will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years old) men or women, hospitalized or not hospitalized, diagnosed for SARS-CoV-2 infection by PCR, with at least one associated risk factor. Considered risk factors are:

   * Age ≥ 65 years
   * Obesity defined as BMI ≥ 30
   * Recent history of uncontrolled High Blood Pressure (SBP > 150 mm Hg DBP >100 mm Hg) according to investigator
   * Treated diabetes (type I or II)
   * History of ischemic cardiovascular disease
2. Symptomatic patients at enrollment. Symptoms are defined as fever (body temperature ≥ 37.8 C oral/tympanic, or ≥ 38.2 C rectal) for more than 24 hours associated either with headache, sore throat, dry cough, fatigue, chest pain or choking sensation (with no associated respiratory distress), myalgia, anosmia or ageusia.
3. Patients with pulse oximetry arterial saturation ≥ 92 % on room air at enrolment.
4. Patients with the following hematological and biochemical laboratory parameters obtained within 7 days prior to Day 0:

   * Hemoglobin above 9.0 g / dL
   * Absolute Neutrophil Count ≥ 1000 / mm3
   * Platelets ≥ 100 000 mm3;
   * Creatinine clearance ≥ 50 mL / min by the Cockcroft Gault formula
   * Total serum bilirubin < 2 x ULN
   * Alkaline phosphatase < 2 x ULN, AST (SGOT) and ALT (SGPT) < 3 x ULN;

Exclusion Criteria:

1. Patients with moderate or severe acute respiratory failure or requiring noninvasive ventilation or oxygen or with SpO2 < 92% or tachypnea (respiratory rate ≥ 30 breaths/min).
2. Patients treated with immunosuppressors and/or immunomodulators.
3. Engrafted patients (organ and/or hematopoietic stem cells).
4. Patients with uncontrolled auto-immune disease.
5. Patients with known or suspected active (i.e. not controlled) bacterial, viral (excluding COVID-19) or fungal infections.
6. Patients with preexisting, severe and not controlled organ failure.
7. History or active malignancy requiring chemotherapy or radiation therapy (excluding 2 years disease free survivor patients).
8. Pregnant or breast-feeding women.
9. Illicit drug or alcohol abuse or dependence that may compromise the patient's safety or adherence to the study protocol.
10. Use of any investigational or non-registered product within 3 months or within 5 half-lives preceding baseline, whichever is longer.
11. Hypersensitivity to ABX464 and/or its excipients.
12. Any condition, which in the opinion of the investigator, could compromise the patient's safety or adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric CUA, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (30):
- Belgium (3):
  - Centre hospitalier Saint Pierre, Brussels
  - Hôpital Erasme, Brussels
  - UZ Gent, Ghent
- Brazil (5):
  - Fundacao de Medicina Tropical Doutor Heitor Vieira Dourado - Instituto de Pesquisa Clínica Carlos Borborema, Manaus, Amazonas
  - Centro Oncológico de Roraima - CECOR - NAP, Boa Vista, Roraima
  - Hospital das Clinicas da FMUSP, São Paulo, São Paulo
  - Instituto Nacional de Infectologia Evandro Chagas - FIOCRUZ Rio de Janeiro, Rio de Janeiro
  - Conjunto Hospitalar do Mandaqui, São Paulo
- France (4):
  - Hôpital Nord, Amiens
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital Saint-Antoine, Paris
- Germany (4):
  - Universitätsmedizin Mannheim Ruprecht-Karls-Universität Heid, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Klinik Altona, Hamburg
- Italy (6):
  - Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico - Infectious Diseases, Milan, Lombardy
  - Ospedale San Paolo, Milan, Lombardy
  - Ospedale Luigi Sacco, AO-PU, Milan, Lombardy
  - Ospedale di Vittorio Veneto - Medecina generale, Vittorio Veneto, Treviso
  - Ospedale A. Manzonidi Lecco - ASST Lecco, Lecco
  - Ospedale Niguarda, Milan
- Mexico (2):
  - Consultorio médico, Mérida, Yucatán
  - Centro de Prevención y Rehabilitación de Enfermedades Pulmon, Nuevo León
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - H.G.U. Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital de La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ABX464: ABX464 50 mg once a day (oral capsule) for 28 days + Standard of Care (SOC)
- Placebo: Placebo 50 mg once a day (oral capsule) + Standard of Care (SOC)
Period: Overall Study
Arm/Group | ABX464 | Placebo
Started | 339 | 170
Completed | 188 | 99
Not Completed | 151 | 71
Not completed — Adverse Event | 11 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 6 | 4
Not completed — Withdrawal by Subject | 24 | 8
Not completed — Lost to Follow-up | 5 | 4
Not completed — Other reasons+ trial site terminated by sponsor + Study terminated by sponsor | 94 | 49
Not completed — End of Study date not collected in the eCRF | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABX464 | Placebo | Total
Number analyzed (Participants) | 339 | 170 | 509
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 240 | 120 | 360
  >=65 years | 98 | 50 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (15.36) | 54.4 (15.05) | 54.7 (15.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 84 | 244
  Male | 179 | 86 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 274 | 130 | 404
  Not Hispanic or Latino | 54 | 35 | 89
  Unknown or Not Reported | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  Belgium | 2 | 2 | 4
  Brazil | 238 | 114 | 352
  Italy | 20 | 11 | 31
  Mexico | 8 | 7 | 15
  United Kingdom | 1 | 0 | 1
  Germany | 2 | 2 | 4
  Spain | 24 | 15 | 39
  France | 20 | 12 | 32
  Peru | 24 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Rate of Responders: i.e. Rate of Patients Who do Not Require Use of High-flow Oxygen Invasive or Non-invasive Mechanical Ventilation (IMV and NIV, Respectively) Within 28 Days and Who Are Alive at the End of the 28 Days Period.
Description: Subjects will be assessed as responders if they did not receive oxygen supplementation through IMV and NIV during the treatment period, and they are alive at the end of the 28-days treatment period.
  Non responders are subjects who receive oxygen supplementation (through IMV and NIV during the treatment period) and/or who die during the 28-days treatment period.
  The use of high-flow oxygen being defined as settings of 3 L/min or greater AND with at least one SpO2 measurement < 92%, with or without O2 supplementation). Descriptive statistics will be presented by treatment arm.
Time Frame: 28 days
Population: An interim analysis was triggered when the first 305 patients were randomized in the study. Randomization was not discontinued during the interim analysis. As the study was stopped for futility based on the interim analysis results, no efficacy data were collected for the patients who were randomized but not included in the interim analysis. Efficacy results are only available for the 305 patients randomized at the time of the interim analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 203 | 102
Participants
  Responder | 169 | 87
  Non-responder | 24 | 7
  Missing | 10 | 8

2. Secondary Outcome: Rate of Patients Hospitalized
Description: To evaluate the proportion of patients requiring hospitalization during the study compared to the {Standard of Care + placebo} group An interim analysis was triggered when the first 305 patients were randomized in the study. As the study was stopped for futility based on the interim analysis results, no efficacy data were collected for the patients who were randomized but not included in the interim analysis. Efficacy results are only available for the 305 patients randomized at the time of the interim analysis.
Time Frame: 28 days
Population: Number of patients randomized at time of Interim analysis
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 203 | 102
Participants | 23 | 11

3. Secondary Outcome: Percentage of Patients Reporting Each Severity Rating on a 7-point Ordinal Scale
Description: 7-point ordinal scale is defined as Not hospitalized, no limitations on activities; Not hospitalized, limitation on activities; Hospitalized, not requiring supplemental oxygen; Hospitalized, requiring supplemental oxygen; Hospitalized, on non-invasive ventilation or high flow oxygen devices; Hospitalized, on invasive mechanical ventilation or ECMO; Death
  An interim analysis was triggered when the first 305 patients were randomized in the study. As the study was stopped for futility based on the interim analysis results, no efficacy data were collected for the patients who were randomized but not included in the interim analysis. Only key outcome analysis was performed during this interim analysis. After discontinuation of the study for futility, Abivax decided to not perform the analysis on this secondary outcome (SAP was amended accordingly). Therefore, these data are not available.
Time Frame: 28-day treatment period
Population: Analysis not done at time of interim analysis. After discontinuation of the study for futility, no further efficacy analysis were done
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Enrolment in Inflammatory Markers in Plasma and in Immune Phenotype and Assessment of Cell-activation Markers in PBMCs
Description: An interim analysis was triggered when the first 305 patients were randomized in the study. As the study was stopped for futility based on the interim analysis results, no efficacy data were collected for the patients who were randomized but not included in the interim analysis. Only key outcome analysis was performed during this interim analysis. After discontinuation of the study for futility, Abivax decided to not perform the analysis on this secondary outcome (SAP was amended accordingly). Therefore, these data are not available.
Time Frame: at each study visit during the 28-day treatment period
Population: as for outcome 3
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Rate of Patients Requiring Oxygen Supplementation
Description: as for outcome 4
Time Frame: 28-day treatment period
Population: as for outcome 3
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Hospitalization
Description: as for outcome 4
Time Frame: 28-day treatment period
Population: as for outcome 3
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Assisted Ventilation and Oxygen Supplementation
Description: as for outcome 4
Time Frame: 28-day treatment period
Population: as for outcome 3
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in microRNA-124 Levels
Description: as for outcome 4
Time Frame: at each study visit during the 28-day treatment period
Population: as for outcome 3
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in CRP, Troponin I & T and D-dimer
Description: as for outcome 4
Time Frame: at each study visit during the 28-day treatment period
Population: as for outcome 3
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: SARS-CoV-2 Viral Load
Description: Nasopharyngeal sample and/or in blood
  An interim analysis was triggered when the first 305 patients were randomized in the study. As the study was stopped for futility based on the interim analysis results, no efficacy data were collected for the patients who were randomized but not included in the interim analysis. Only key outcome analysis was performed during this interim analysis. After discontinuation of the study for futility, Abivax decided to not perform the analysis on this secondary outcome (SAP was amended accordingly). Therefore, these data are not available.
Time Frame: at each study visit during the 28-day treatment period
Population: as for outcome 3
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number and Rates of Participants With Treatment Emergent Adverse Event
Description: Number and rates of participants included in the safety analysis set who had Treatment Emergent Adverse Event
Time Frame: From D0 to D48 (28 days treatment period + up to 20 days Safety follow-up period)
Population: Analysis of safety was performed on the safety data set consisting in all patients who received at least one dose of ABX464 in the study. A total of 505 patients were included in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 | Placebo
Number analyzed (Participants) | 335 | 170
Participants
  Period 1: AE onset or worsens before or on Day 28 | 209 | 83
  Period 2: AE onset or worsens after Day 28 | 22 | 20

ADVERSE EVENTS:
Time Frame: 49 days
Arm/Group | ABX464 | Placebo
All-Cause Mortality (participants affected / at risk) | 6/335 | 4/170
Serious Adverse Events (participants affected / at risk) | 36/335 | 20/170
Other Adverse Events (participants affected / at risk) | 115/335 | 27/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 (N=335) | Placebo (N=170)
covid-19 (Infections and infestations) | 10 (10) | 2 (2)
Covid-19 pneumonia (Infections and infestations) | 5 (5) | 5 (5)
Severe acute respiratory syndrome (Infections and infestations) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrintestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 2 (2)
Hepatic artery embolism (Hepatobiliary disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 (N=335) | Placebo (N=170)
Abdominal pain upper (Gastrointestinal disorders) | 32 (34) | 5 (5)
Diiarrhoea (Gastrointestinal disorders) | 30 (31) | 6 (6)
Nausea (Gastrointestinal disorders) | 20 (21) | 6 (7)
Headache (Nervous system disorders) | 49 (51) | 19 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (24) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT04393038/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04393038/SAP_001.pdf